CLINICAL TRIAL: NCT04633278
Title: A Multicenter, Phase 2, Open-label Study of Intratumoral CMP-001 in Combination With Intravenous Pembrolizumab in Subjects With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: CMP-001 in Combination With Pembrolizumab in Subjects With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decision
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMP-001-007
Record Dates: First submitted 2020-10-26; First posted 2020-11-18 (Actual); Results first posted 2025-04-08 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Head and Neck Cancer; Pembrolizumab; Carcinoma; HNSCC
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CMP-001 and Pembrolizumab (Experimental): All subjects will receive CMP-001 IT and pembrolizumab IV according to the treatment schedule until a reason for treatment discontinuation is reached.
  Interventions: Drug: CMP-001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CMP-001 — Subjects will receive CMP-001 10mg weekly for 2 doses after which CMP-001 will be administered every 3 weeks. The first dose of CMP-001 may be administered subcutaneously (SC) or Intratumorally (IT) at the discretion of Investigator. All subsequent doses will be injected intratumorally every 3 weeks (Q3W).
  Other Names: vidutolimod
Drug: Pembrolizumab — Pembrolizumab 200 mg IV is administered Q3W.
  Other Names: Keytruda

SUMMARY:
CMP-001-007 is a Phase 2 study of CMP-001 intratumoral (IT) and pembrolizumab intravenous (IV) administered to participants with head and neck squamous cell carcinoma (HNSCC) who have not been previously treated with a programmed cell death protein 1 (PD-1) blocking antibody.

The primary objective of the study is to determine the Investigator-assessed confirmed objective response with CMP-001 in combination with pembrolizumab in subjects with head and neck squamous cell carcinoma (HNSCC)

The secondary objectives are to:

* To evaluate the safety and tolerability of CMP-001 administered by intratumoral (IT) injection in combination with pembrolizumab in subjects with HNSCC
* To evaluate the efficacy of CMP-001 in combination with pembrolizumab in subjects with HNSCC
* To evaluate the effect of human papillomavirus (HPV) infection and programmed death-ligand 1 (PD-L1) expressions on the efficacy of CMP-001 in combination with pembrolizumab

Participants will continue to receive treatment of CMP-001 and pembrolizumab according to the treatment schedule until a reason for treatment discontinuation is reached.

DETAILED DESCRIPTION:
Former Sponsor Checkmate Pharmaceuticals

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically-confirmed recurrent or metastatic HNSCC considered incurable by local therapies.
* No prior systemic therapy in the recurrent or metastatic setting. Systemic therapy as part of multi-modal treatment for locally advanced disease is allowed.
* Primary tumor locations of oropharynx, oral cavity, hypopharynx, larynx or paranasal sinus. Participants may not have a primary tumor site of nasopharynx (any histology).
* Able to provide tissue from a core or excisional biopsy (fine needle aspirate is not sufficient). A newly obtained biopsy (within 90 days before the start of study treatment) is preferred but an archival sample is acceptable.
* Combined Positive Score (CPS) ≥ 1 for PD-L1 on Immunohistochemistry (IHC) of tumor tissue.
* Have results of tumor HPV p16 by IHC for oropharyngeal cancer.
* Measurable disease as defined by RECIST v1.1, and both of the following:

  1. At least 1 lesion amenable to repeated Intratumoral (IT) injection.
  2. Documented disease progression in any lesion that was previously radiated in order to serve as a target lesion.
* Adequate organ function based on most recent laboratory values within 3 weeks before the first dose of study drug on Week 1 Day 1 (W1D1) Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1 at Screening.
* Capable of understanding and complying with protocol requirements.
* Women of childbearing potential must have negative serum pregnancy test during Screening and be willing to use an adequate method of contraception from the time of consent until at least 120 days after the last dose of study drug.
* Male subjects must be surgically sterile or must agree to use adequate method of contraception from the time of consent until at least 120 days after the last dose of study drug.
* Able and willing to provide written informed consent and to follow study instructions.
* Subjects unable to provide written informed consent on their own behalf will not be eligible for the study.

Exclusion Criteria:

* Disease suitable for local therapy administered with curative intent.
* Has PD within 3 months of completion of curatively intent systemic treatment for locoregionally advanced HNSCC.
* Radiation therapy (or other non-systemic therapy) within 2 weeks before the first dose of study drug on W1D1.
* Received prior therapy with PD-1 or PD-L1 blocking antibody therapy in the recurrent/ metastatic setting. If PD-1 or PD-L1 blocking antibody therapy was given as part of curative intent therapy, it must be at least 1 year since receipt of PD-1 or PD-L1 blocking antibody.
* Not fully recovered from adverse events (to Grade 1 or less [per CTCAE v5.0]), with the exception of persistent alopecia, neuropathy, ototoxicity, hypothyroidism, pain, or dysphagia, due to prior treatment.
* Requires systemic pharmacologic doses of corticosteroids greater than the equivalent of 10 mg/day prednisone within 30 days before the first dose of study drug on W1D1.

  1. Subjects who are currently receiving steroids at a prednisone-equivalent dose of ≤ 10 mg/day do not need to discontinue steroids prior to enrollment.
  2. Replacement doses, topical, ophthalmologic, and inhalational steroids are permitted.
* Active pneumonitis, history of noninfectious pneumonitis that required steroids, or history of interstitial lung disease.
* Severe uncontrolled cardiac disease within 6 months of Screening, including but not limited to poorly controlled hypertension, unstable angina, myocardial infarction, congestive heart failure (New York Heart Association Class II or greater), pericarditis within the previous 6 months, cerebrovascular accident, implanted or continuous use of a pacemaker or defibrillator.
* Known history of immunodeficiency.
* Known additional malignancy that is progressing or required active treatment within the past 3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, curatively treated localized prostate cancer with non-detectable prostate-specific antigen, in situ cervical cancer on biopsy or a squamous intraepithelial lesion on Papanicolaou smear, and thyroid cancer (except anaplastic).
* Active autoimmune disease that has required systemic treatment in past 2 years; replacement therapy is not considered a form of systemic treatment
* Untreated, symptomatic, or enlarging central nervous system (CNS) metastases or carcinomatous meningitis.
* Prior allogenic tissue/solid organ transplant.
* Active infection requiring systemic therapy.
* Known or suspected active infection with SARS-CoV-2 virus.
* Known or suspected infection with human immunodeficiency virus, hepatitis B virus or hepatitis C virus; testing is not required unless suspected.
* Received a live virus vaccination within 30 days before the start of study drug dosing on W1D1.
* Received blood products (including platelets or red blood cells) or colony stimulating factors [including granulocyte colony-stimulating factor (GCSF), granulocyte-macrophage colony-stimulating factor (GMCSF) (or recombinant erythropoietin)] within 30 days before the start of Screening.
* Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the Investigator, would make the subject unable to cooperate or participate in the trial.
* Participation in another clinical trial of an investigational anticancer therapy or device within 30 days before the first dose of study drug.
* Requires prohibited treatment (ie. non-protocol specified anticancer pharmacotherapy, surgery or conventional radiotherapy for treatment of malignant tumor).
* Has a life expectancy of less than 3 months and/or has rapidly progressing disease (eg. tumor bleeding, uncontrolled tumor pain) in the opinion of the treating Investigator.
* Received previous CMP-001 treatment.
* Pregnant or breast-feeding or expecting to conceive or father children within the projected duration of the study, from the time of consent until at least 120 days after the last dose of study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (19):
- United States (19):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California - San Diego, La Jolla, California
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Hematology-Oncology, Los Angeles, California
  - University of Southern California: Norris Oncology/Hematology - Newport Beach, Newport Beach, California
  - University Cancer & Blood Center, Athens, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Atlantic Health, Morristown, New Jersey
  - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - UPMC - Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Bon Secours St. Francis Cancer Center, Greenville, South Carolina
  - University of Tennessee, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital/Cancer Center, Houston, Texas
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Groups:
- CMP-001 IT + Pembrolizumab - Schedule A: Participants received CMP-001 intratumorally (IT) and pembrolizumab intravenously (IV) according to treatment schedule A.
- CMP-001 IT + Pembrolizumab - Schedule B: Participants received CMP-001 IT and pembrolizumab IV according to treatment schedule B.
Period: Overall Study
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Started (Received at least 1 dose of study treatment) | 17 | 7
Completed | 0 | 0
Not Completed | 17 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 11 | 7
Not completed — Sponsor Decision | 3 | 0
Not completed — Not Listed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B | Total
Number analyzed (Participants) | 17 | 7 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.1 (8.57) | 71.0 (10.33) | 66.1 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 13 | 4 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 7 | 22
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 15 | 7 | 22
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Confirmed Objective Response Rate (ORR)
Description: Confirmed ORR is defined as the percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as determined by Investigator assessment (IA).
Time Frame: Up to approximately 109 weeks
Population: Treated Analysis Set (All participants who received at least 1 dose of CMP-001)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 17 | 7
Percentage of participants | 17.6 [3.80 to 43.43] | 0 [0.00 to 40.96]

2. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE), Any Serious TEAE, and Any TEAE Leading to Discontinuation or Death
Description: TEAE is defined as an AE that started or worsened in severity on or after the date that study drug was first administered (W1D1) until 30 days after the last dose of study treatment.
Time Frame: Up to approximately 109 weeks
Population: Treated Analysis Set (All participants who received at least 1 dose of CMP-001)
Measure: Number; unit: Participants
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 17 | 7
Participants
  Any TEAE | 17 | 7
  Any serious TEAE | 7 | 5
  Any TEAE leading to death | 1 | 0

3. Secondary Outcome: Severity of TEAEs as Assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 5.0
Description: NI CTCAE Adverse Event Grades:
  Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated Grade 2 Moderate; minimal, local, or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limited self-care activities of daily living Grade 4 Life-threatening consequences: urgent intervention indicated Grade 5 Death related to adverse event
Time Frame: Up to approximately 109 weeks
Population: Treated Analysis Set (All participants who received at least 1 dose of CMP-001)
Measure: Number; unit: Participants
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 17 | 7
Participants
  Grade 1 - 2 | 7 | 1
  Grade 3 | 7 | 6
  Grade 4 | 2 | 0
  Grade 5 | 1 | 0

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR, defined as the time from date of first documented response (CR or PR) to date of documented PD, based on RECIST v1.1 by Investigator assessment (IA).
Time Frame: Up to approximately 28 months (120 weeks)
Population: Number of participants analyzed for DOR includes only participants who have a confirmed best overall response (BOR) of complete response (CR) or partial response (PR).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 3 | 0
Months | NA [2.825 to NA] — Not evaluable due to low number of participants analyzed. |

5. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: Progression-free Survival (PFS), defined as the time from date of first dose of study drug to date of documented PD based on RECIST v1.1 by IA or death, whichever occurs first.
Time Frame: Up to approximately 28 months (120 weeks)
Population: Treated Analysis Set (All participants who received at least 1 dose of CMP-001)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 17 | 7
Months | 2.103 [1.183 to 6.472] | 1.807 [1.478 to 3.450]

6. Secondary Outcome: Duration of Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from the first dose date of the study treatment to the date of death from any cause.
Time Frame: From first dose up to approximately 28 months (120 weeks)
Population: Treated Analysis Set (All participants who received at least 1 dose of CMP-001)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 17 | 7
Months | 6.932 [2.333 to 14.456] | 7.129 [1.643 to 12.287]

7. Secondary Outcome: Immune Objective Response Rate (iORR)
Description: Immune objective response rate (iORR), defined as the percentage of participants who have an immune best overall response (iBOR) of immune complete response (iCR) or immune partial response (iPR) based on the immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) as determined by Investigator.
Time Frame: Up to approximately 109 weeks
Population: Treated Analysis Set (All participants who received at least 1 dose of CMP-001)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 17 | 7
Percentage of participants | 0 [0.00 to 97.50] | 0 [0.00 to 84.19]

8. Secondary Outcome: Immune Progression-free Survival (iPFS)
Description: iPFS, defined as the time from date of first dose of study drug to date of immune Confirmed Progressive Disease (iCPD) based on immunotherapy Response Evaluation Criteria in Solid Tumors (iRECIST) by IA or death, whichever occurs first.
Time Frame: Up to approximately 28 months (120 weeks)
Population: Number analyzed = Number of participants continuing study treatment beyond PD.
Measure: Median (Full Range); unit: Months
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 1 | 2
Months | 9.955 [9.955 to 9.955] | NA [3.38 to 3.45] — Data not available due to insufficient number of participants with events.

9. Secondary Outcome: Confirmed ORR Based on Human Papillomavirus (HPV) Status
Description: Confirmed ORR is defined as the percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as determined by Investigator assessment (IA) based on HPV status.
Time Frame: Up to approximately 109 weeks
Population: Subgroup of participants in Treated Analysis Set that completed HPV testing
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 10 | 6
Percentage of participants
  HPV positive: number analyzed (Participants) | 6 | 1
  HPV positive | 16.7 [0.42 to 64.12] | 0 [0.00 to 97.50]
  HPV negative: number analyzed (Participants) | 4 | 5
  HPV negative | 25.0 [0.63 to 80.59] | 0 [0.00 to 52.18]

10. Secondary Outcome: Confirmed ORR Based on Programmed Death-ligand 1 (PD-L1) Expressions
Description: Confirmed ORR is defined as the percentage of participants with a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as determined by Investigator assessment (IA) based on PD-L1 expressions (combined positive score [CPS] ≥ 1 and CPS ≥ 20)
Time Frame: Up to approximately 109 weeks
Population: Subgroup of participants in Treated Analysis Set that had PL-1 expressions; For 1 participant, the site used a local, qualitative test (positive/negative). Therefore, the CPS (%) is missing for this 1 participant.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 17 | 6
Percentage of participants
  PD-L1 Expression: 1 to < 20: number analyzed (Participants) | 10 | 2
  PD-L1 Expression: 1 to < 20 | 20.0 [2.52 to 55.61] | 0 [0.00 to 84.19]
  PD-L1 Expression: >= 20: number analyzed (Participants) | 7 | 4
  PD-L1 Expression: >= 20 | 14.3 [0.36 to 57.87] | 0 [0.00 to 60.24]

11. Secondary Outcome: Duration of PFS Based on HPV Status
Description: Progression-free Survival (PFS), defined as the time from date of first dose of study drug to date of documented PD based on RECIST v1.1 by IA or death, whichever occurs first. PFS based on HPV status
Time Frame: Up to approximately 28 months (120 weeks)
Population: Subgroup of participants in Treated Analysis Set that completed HPV testing
Measure: Median (Full Range); unit: Months
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 10 | 6
Months
  HPV positive: number analyzed (Participants) | 6 | 1
  HPV positive | 3.253 [0.72 to 22.44] | 3.975 [3.975 to 3.975]
  HPV negative: number analyzed (Participants) | 4 | 5
  HPV negative | 1.183 [0.03 to 6.90] | 1.807 [1.48 to 3.45]

12. Secondary Outcome: Immune Duration of Response (iDOR)
Description: iDOR, defined as the time from the date of the first immune response (iCR or iPR) to the date of immune confirmed progressive disease (iCPD) by IA.
Time Frame: Up to approximately 28 months (120 weeks)
Population: Number analyzed = Number of participants who had iBOR of immune complete response (iCR) or immune partial response (iPR). Here, 0 participants met the criteria.
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: DOR Based on HPV Status
Description: DOR, defined as the time from date of first documented response (CR or PR) to date of documented PD, based on RECIST v1.1 by Investigator assessment (IA). DOR based on HPV status.
Time Frame: Up to approximately 28 months (120 weeks)
Population: Number of participants analyzed for DOR based on HPV status includes only participants who have a confirmed best overall response (BOR) of complete response (CR) or partial response (PR) to date of documented PD and completed HPV testing.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 2 | 0
Months
  HPV negative: number analyzed (Participants) | 1 | 0
  HPV negative | NA [NA to NA] — Data not available due to insufficient number of participants with events. |
  HPV positive: number analyzed (Participants) | 1 | 0
  HPV positive | NA [NA to NA] — Data not available due to insufficient number of participants with events. |

14. Secondary Outcome: DOR Based on PD-L1 Expressions
Description: DOR, defined as the time from date of first documented response (CR or PR) to date of documented PD, based on RECIST v1.1 by Investigator assessment (IA). DOR based on PD-L1 expressions (combined positive score [CPS] 20).
Time Frame: Up to approximately 28 months (120 weeks)
Population: Number of participants analyzed for DOR based on PD-L1 expressions included only participants with confirmed BOR of CR or PR and CPS >=20. Here, 0 participants met the criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 1 | 0
Months | NA [NA to NA] — Data not available due to insufficient number of participants with events. |

15. Secondary Outcome: PFS Based on PD-L1 Expressions
Description: Progression-free Survival (PFS), defined as the time from date of first dose of study drug to date of documented PD based on RECIST v1.1 by IA or death, whichever occurs first. PFS based on PD-L1 expressions (combined positive score [CPS] 20).
Time Frame: Up to approximately 28 months (120 weeks)
Population: Number of participants analyzed for PFS based on PD-L1 expressions included only participants with documented PD or death and CPS >=20. Here, 0 participants met the criteria.
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From signing of informed consent through end of study up to approximately 28 months (120 weeks)
Arm/Group | CMP-001 IT + Pembrolizumab - Schedule A | CMP-001 IT + Pembrolizumab - Schedule B
All-Cause Mortality (participants affected / at risk) | 11/17 | 7/7
Serious Adverse Events (participants affected / at risk) | 7/17 | 5/7
Other Adverse Events (participants affected / at risk) | 17/17 | 6/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMP-001 IT + Pembrolizumab - Schedule A (N=17) | CMP-001 IT + Pembrolizumab - Schedule B (N=7)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Bacterial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMP-001 IT + Pembrolizumab - Schedule A (N=17) | CMP-001 IT + Pembrolizumab - Schedule B (N=7)
Chills (General disorders) | 8 (8) | 3 (4)
Pyrexia (General disorders) | 7 (8) | 1 (2)
Fatigue (General disorders) | 3 (3) | 2 (2)
Injection site pain (General disorders) | 3 (9) | 0 (0)
Facial pain (General disorders) | 2 (3) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1)
Injection site oedema (General disorders) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 1 (1) | 0 (0)
Injection site vesicles (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (2) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 5 (7) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (5) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 3 (5) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (3) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral lichen planus (Gastrointestinal disorders) | 1 (2) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (5) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 2 (2)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic hypertension (Vascular disorders) | 1 (2) | 0 (0)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (4) | 0 (0)
Muscle discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 3 (3) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 2 (3) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (2) | 0 (0)
Blood pressure diastolic decreased (Investigations) | 1 (2) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (3)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Procalcitonin increased (Investigations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tumour fistulisation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (3) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injection related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Ear discomfort (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
Per sponsor's decision, enrollment was stopped before reaching the full sample size as originally planned for the analyses described in the protocol. This was a development decision independent of the safety or efficacy profile/findings associated with the study. All analyses are hence exploratory. The performance of the statistical analysis for the protocol objectives and endpoints of the exploratory phase 2 study is limited by the limited availability of the data source.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the Sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2024-11-21): https://cdn.clinicaltrials.gov/large-docs/78/NCT04633278/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT04633278/SAP_001.pdf